CLINICAL TRIAL: NCT04959942
Title: Efficacy of Adding Scapular Stabilization Exercises to Postural Correctional Exercises on Endurance of Cervical Flexor and Extensor Muscles on Asymptomatic Forward Head Posture; Randomized Controlled Trial
Brief Title: Efficacy of Adding Scapular Stabilization Exercises to Postural Correctional Exercises on on Forward Head Posture
Acronym: FHP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Al Shaymaa Shaaban Abd El Azeim, principle investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: p.t.REC/012/003244
Record Dates: First submitted 2021-07-02; First posted 2021-07-13 (Actual); Last update posted 2021-07-13 (Actual); Status verified 2021-07

CONDITIONS: Forward Head Posture
Keywords: scapular stabilization exercise; postural correction exercises; forward head posture
MeSH Terms: interventions — Counseling

STUDY DESIGN:
Intervention Model Description: scapular stabilization and postural correction exercise
Who Masked: Participant, Outcomes Assessor
Masking Description: random generator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- scapular stabilization exercise (Experimental): the subjects will receive scapular stabilization exercise + postural correction exercise and advice three times per week for 10 weeks
  Interventions: Other: scapular stabilization exercise
- postural correction exercise (Experimental): the subjects will receive postural correction exercise and advice three times per week for 10 weeks
  Interventions: Other: scapular stabilization exercise; Other: postural correction exercise
- advice (Active Comparator): the subjects will receive advice three times per week for 10 weeks
  Interventions: Other: scapular stabilization exercise; Other: postural correction exercise; Other: advice

INTERVENTIONS:
Other: scapular stabilization exercise — In the supine position, the subject will instruct to take a deep breath to relax the body. In croock-lying position, the subject will raise his dominant arm to 90° shoulder flexion with full elbow extension and scapular protraction. In the quadruped position, the subject lifts up his arms alternatively with shoulder abduction and 120 ° flexion. In a sitting position with 90° knee flexion on a stool or bed without back support, the subject held a pair of dumbbells (2 kg) in each hand and laterally lifted them up while maintaining the height of scapulae below 80°. Each stage will instruct to be held for 10 seconds before returning to the starting position and three laps of 10 repetitions with a 30-second break in between will perform. In the sitting position, a mirror will place in front of the patient. The subject will instruct to check and correct his posture by him
Other: postural correction exercise — The program consisted of two strengthening (deep cervical flexors and scapular retractors) and two stretchings: cervical extensors (sub-occipital muscles) and pectoral muscles). The program was based on a program by Harman and Kendall.
  Arms: advice; postural correction exercise
Other: advice — all subjects will be instructed to maintain normal alignment of the cervical vertebry
  Arms: advice

SUMMARY:
The aim of this study is to investigate efficacy of adding Scapular Stabilization Exercises to postural correctional exercises on Endurance of cervical flexor and extensor muscles on Asymptomatic forward head posture.

DETAILED DESCRIPTION:
Forward head posture (FHP) is the most common deviation from ideal head posture and is characterized by the head projecting forward into the sagittal plane such that it is anterior to the trunk. Individuals with neck pain frequently demonstrate FHP, when compared to age-matched controls.

Asymmetric posture is a chronic stressor and the origin of most noxious stimuli that could alleviate 70-90 % of chronic pain. It is reported that FHP is a common postural abnormality, with a conservative estimate being 66 % of the patient population. It causes vertebral displacement patterns, abnormal stresses, and strain on the spinal cord. FHP has adverse mechanical tension on neural and vascular elements.

It is theorized that when muscle performance is impaired, the balance between the stabilizers on the posterior aspect of the neck and the DNFs will be disrupted, resulting in loss of proper alignment and posture, which is then likely to contribute to cervical Impairment (loss of range of motion, or decreased strength including, but not limited to, the sternocleidomastoid (SCM), trapezius, and deep neck flexor (DNF) muscles endurance of the neck musculature.

Assessment of DNF muscle performance properties is arguably important given the relationship between DNF muscle torque and endurance deficits and patient complaints of head and neck pain. sixty subjects with forward head posture assigned randomly to three groups. experimental group 1 will receive scapular stabilization plus postural correction exercise and advice, experimental group 2 will receive postural correction exercise plus advice and finally control group will receive advice.

ELIGIBILITY:
Inclusion Criteria:

1. If asymptomatic subjects with CVA equal or less than 50.
2. shoulder flexion at least 130 degrees or more, they involved in this research.

Exclusion Criteria:

1. If they had a history of cervical spine sur¬gery
2. Cervical spondylosis
3. Cervical or shoulder neurological movement disorder, Temporo-mandibular surgery, Pathologic trauma.

Ages: 20 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-07-15 (Estimated); Primary Completion 2021-09-30 (Estimated); Study Completion 2021-09-30 (Estimated)

PRIMARY OUTCOMES:
craniovertebral angle | up to ten weeks
  craniovertebral angle will be measured by objective software.
cervical range of motion | up to ten weeks
  cervical range of motion will be assessed by CROM. cervical flexion, extension, side bending and rotation will be assessed

SECONDARY OUTCOMES:
flexion endurance | up to ten weeks
  flexion endurance test by stop watch will be used for assessment the endurance of cervical flexor
extension endurance | up to ten weeks
  extension endurance test by stop watch will be used for assessment the endurance of extensor muscles
muscle activity during rest and activity | up to ten weeks
  electromyography will be used for measuring the activity of upper trapezius and sternocleidomastoid muscle at rest and during activity